CLINICAL TRIAL: NCT04261712
Title: An Open Label, Long-term Extension Study to Evaluate the Safety and Efficacy of CRN00808 in Subjects With Acromegaly (ACROBAT Advance)
Brief Title: A Study to Evaluate the Long-Term Safety and Efficacy of Paltusotine for the Treatment of Acromegaly (ACROBAT Advance)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRN00808-05; U1111-1245-5276 (Other: WHO); 2019-002193-31 (EudraCT Number); 2024-511921-75-00 (EU CTIS Number)
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acromegaly
Keywords: Acromegaly; ACROBAT; ADVANCE; Paltusotine
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Paltusotine (Experimental)
  Interventions: Drug: Paltusotine

INTERVENTIONS:
Drug: Paltusotine — Paltusotine, once daily by mouth
  Other Names: CRN00808

SUMMARY:
A phase 2, open label, long-term extension study designed to evaluate the safety and efficacy of paltusotine (formerly CRN00808; an oral selective nonpeptide somatostatin receptor type 2 biased agonist) in subjects with acromegaly.

ELIGIBILITY:
Inclusion Criteria:

1. Completed one of the parent studies (Acrobat Evolve [CRN00808-02] or Acrobat Edge [CRN00808-03])
2. Females must be non-pregnant and non-lactating, and either surgically sterile, post-menopausal, or using effective method(s) of birth control
3. Willing to provide signed informed consent

Exclusion Criteria:

1. Clinically significant concomitant disease including, but not limited to, cardiovascular disease; moderate or severe renal insufficiency; or significant liver disease (including cirrhosis)
2. Pituitary radiation since completing participation in parent studies
3. History or presence of malignancy except adequately treated basal cell and squamous cell carcinomas of the skin within the past 5 years
4. Positive test at Screening for HIV, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV-Ab).
5. History of alcohol or substance abuse in the past 12 months
6. Use of any investigational drug (other than paltusotine) within the past 30 days or 5 half-lives, whichever is longer before Screening
7. Any condition that in the opinion of the investigator would jeopardize the subject's appropriate participation in this study.
8. Cardiovascular conditions or medications associated with prolonged QT or those which predispose subjects to heart rhythm abnormalities
9. Subjects with symptomatic cholelithiasis
10. Subjects with clinically significant abnormal findings during the Screening Period, and any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardize the subject's safety or ability to complete the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) throughout the study | Week 316

SECONDARY OUTCOMES:
Change in insulin-like growth factor-1 (IGF-1) level | Week 16, Week 312
Change in growth hormone (GH) level | Week 16, Week 312

CONTACTS AND LOCATIONS:
Locations (18):
- United States (6):
  - Crinetics Study Site, Los Angeles, California
  - Crinetics Study Site, Chicago, Illinois
  - Crinetics Study Site, Boston, Massachusetts
  - Crinetics Study Site, Columbus, Ohio
  - Crinetics Study Site, Pittsburgh, Pennsylvania
  - Crinetics Study Site, Dallas, Texas
- Brazil (3):
  - Crinetics Study Site, Curitiba, Paraná
  - Crinetics Study Site, Rio de Janeiro
  - Crinetics Study Site, São Paulo
- Greece (4):
  - Crinetics Study Site, Athens
  - Crinetics Study Site 1, Athens
  - Crinetics Study Site 2, Athens
  - Crinetics Study Site, Thessaloniki
- Hungary (2):
  - Crinetics Study Site, Budapest
  - Crinetics Study Site, Pécs
- Crinetics Study Site, Belgrade, Serbia
- United Kingdom (2):
  - Crinetics Study Site, Coventry
  - Crinetics Study Site, Leeds

IPD SHARING:
Plan to Share IPD: No